CLINICAL TRIAL: NCT06756971
Title: Comparison Between Propofol and Dexmedetomidine as Anesthetic Protocols for Drug Induced Sleep Endoscopy (DISE) in Pediatric Patients With Sleep Disordered Breathing: A Prospective Randomized Controlled Trial
Brief Title: DISE in Pediatric Sleep Disordered Breathing
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI moved to another institution
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 202011387
Record Dates: First submitted 2022-05-21; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Sleep Disordered Breathing; Drug Induced Sleep Disorder
Keywords: Drug induced sleep endoscopy; sleep disordered breathing; DISE directed surgery; children
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This study will randomize n=120 study participants undergoing DISE to one of two anesthetic agents, Propofol or Dexmedetomidine. With equal allocation to each arm (n=60 per group).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Once consent is obtained, the patient will be recruited. Name and surgical date will be provided to our statistician. Permuted block randomization will be performed. The patient will either receive Propofol or Dexmedetomidine as the anesthetic regimen intraoperatively. This will be delivered by the anesthesia team. The surgeon will be blinded, so as the patient. The anesthetist will not be blinded. DISE, adenotonsillectomy or DISE directed surgery will be performed. Data will be collected by the research team throughout the procedure and post procedure.
  This project does not involve the evaluation, or testing, of the safety and/or efficacy of a medical device or a new drug.
  This is an interventional study, in which the investigators are randomly assigning subjects to one of the two anesthetics, Propofol or Dexmedetomidine. All patients will have cardiopulmonary monitoring, and intravenous access.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): Arm 1: Propofol
  1. PO Versed (Benzodiazepine) preoperatively
  2. Obtain baseline bispectral index (BIS) monitor
  3. Mask induction with Sevoflurane
  4. Intravenous access
  5. Propofol bolus 0.5-2 mg/kg to start followed by infusion 200-350 mcg/kg/min
  6. Wait around 2 minutes
  7. BIS monitor with Propofol on board
  Interventions: Drug: Propofol
- Dexmedetomidine (Active Comparator): Arm 2: Dexmedetomidine
  1. PO Versed (Benzodiazepine) preoperatively
  2. Obtain baseline BIS monitor
  3. Mask induction with Sevoflurane
  4. Intravenous access
  5. Dexmedetomidine bolus 0.5-3 mcg/kg to start followed by infusion 0.5-2mcg/kg/hr
  6. Wait around 10 mins
  7. BIS monitor with Dexmedetomidine on board
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol — Propofol will be administered until the patients is in an optimal plane that mimics natural sleep while spontaneously breathing to allow for a DISE evaluation
  Other Names: Diprivan; Fresenius Propoven; Propofol-Lipuro; Propofol-II [DSC]; TEVA-Propofol
  Arms: Propofol
Drug: Dexmedetomidine — Dexmedetomidine will be administered until the patients is in an optimal plane that mimics natural sleep while spontaneously breathing to allow for a DISE evaluation
  Other Names: Precedex
  Arms: Dexmedetomidine

SUMMARY:
Adenotonsillar hypertrophy is the most common reason for children to have sleep disordered breathing (SDB). Even though adenotonsillectomy improves sleep apnea in children, 20-40% of children will still have persistent SDB. Drug Induced Sleep Endoscopy (DISE) is a tool that dynamically evaluates the upper airway during simulated sleep. It identifies sites of upper airway obstruction and/or collapse. It is used to predict which children will get better if their tonsils and adenoids are removed, and which children have other reasons for SDB. DISE is done during a state of simulated sleep. Different anesthetic medications are currently being used. However, there is no identified ideal anesthetic medication to simulate natural sleep. Propofol and Dexmedetomidine are the most frequently used, either alone or in combination with other medications. The aim is to perform a head-to-head study comparing those 2 commonly used regimens. The investigator would like to learn how the anesthetic medication affects performing the procedure and how well our patients tolerate it. This helps us identify an ideal regimen that can be a standardized DISE protocol in the pediatric population in the future. Our objective is to determine which anesthetic regimen, Dexmedetomidine or Propofol, is safer and more efficacious. This will be a randomized controlled trial at the University of Iowa Stead Family Children's Hospital. Children with sleep disordered breathing will undergo DISE and subsequent surgical procedure based on the level of obstruction found during DISE. Via randomization the child will be preselected to have a specific anesthetic for the procedure, either Dexmedetomidine or Propofol. The investigator will record information related to the medications used, the vital signs, the ability to perform DISE fully, the findings seen on DISE and the surgery performed. Consent will be obtained from the legal guardian or parent with legal authority to consent.

DETAILED DESCRIPTION:
Drug-induced sleep endoscopy (DISE) in children has gained popularity in the past 10 years. Its most valuable use is in patients with sleep disordered breathing (SDB). DISE is capable of identifying dynamic sites of upper airway obstruction and or collapse during sleep, beyond the tonsils and adenoids. It is also capable of identifying the degree of dynamic obstruction caused by different anatomical structures. Currently, pediatric patients with SDB diagnosed either clinically with the help of a validated sleep questionnaire or on the basis of sleep study and undergo surgery depending on the level of the obstruction. The surgery most commonly performed is adenotonsillectomy. In order to diagnose the level of obstruction DISE is performed. Currently, there is a lack in consensus regarding the ideal anesthetic regimen to simulate natural sleep and poor agreement regarding DISE anesthetic protocols among experts. An ideal agent would provide sufficient analgesia under near-physiologic settings and prevent substantial airway collapse, respiratory depression, and cardiovascular effects. It should have a predictable period of action and a smooth emergence. Multiple anesthetic regimens have been used for DISE. This includes inhalation anesthesia such as Sevoflurane, total intravenous anesthesia (TIVA) such as Propofol alone or with Remifentanil, and Dexmedetomidine alone or with Ketamine. Propofol and Dexmedetomidine are the most frequently used regimens, either alone or in combination with another medication. Most studies in this regard are retrospective in nature, with only a handful of prospective studies. To date, no randomized controlled trials have been performed to address anesthetic regimens to perform DISE in children. One randomized controlled trial in adults compared Propofol and Dexmedetomidine as anesthetic regimens for DISE and concluded that Dexmedetomidine could satisfy the DISE requirement and had no significant side effects on cardiovascular changes and less interference of breathing. Given the difference between children and adults in pathophysiology, risk factors for the diseases and tolerance of medication, the findings cannot be claimed to be similar in children unless proven. The aim is to perform a head-to-head study comparing the 2 commonly used regimens Propofol and Dexmedetomidine in children with SDB. This helps us identify a safer and more efficacious regimen that can be a standardized DISE protocol in the pediatric population in the future.

ELIGIBILITY:
Inclusion Criteria:

* Children 1 month-18 years of age
* Clinical diagnosis of sleep disordered breathing (SDB) either based on a Pediatric sleep questionnaire (>33% on modified Pediatric Sleep Questionnaire (PSQ)) or Sleep study
* Subject is deemed a surgical candidate for undergoing DISE, adenotonsillectomy or DISE directed surgery

Exclusion Criteria:

* Adult patients
* Hypersensitivity to propofol or dexmedetomidine or any of their components,
* Allergies to eggs, egg products, soybeans, or soy products,
* Congenital cardiac disease, cardiac conduction system pathology, and increased pulmonary artery pressure or decreased cardiac output (e.g., right-sided heart failure, septic shock).
* Children who are receiving medicines with rate-slowing action on the atrioventricular node (eg, digoxin, nifedipine)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Comparing Dexmedetomidine and Propofol for successful DISE (Drug Induced Sleep Endoscopy) procedure in-terms regarding which drug works better without causing side effects | 5-20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sohit Kanotra, MD, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman NR, Parikh SR, Ishman SL, Ruiz AG, El-Hakim H, Ulualp SO, Wootten CT, Koltai PJ, Chan DK. The current state of pediatric drug-induced sleep endoscopy. Laryngoscope. 2017 Jan;127(1):266-272. doi: 10.1002/lary.26091. Epub 2016 Jun 16. PMID 27311407
- [Background] Liu KA, Liu CC, Alex G, Szmuk P, Mitchell RB. Anesthetic management of children undergoing drug-induced sleep endoscopy: A retrospective review. Int J Pediatr Otorhinolaryngol. 2020 Dec;139:110440. doi: 10.1016/j.ijporl.2020.110440. Epub 2020 Oct 14. PMID 33080472
- [Background] Zhao LL, Liu H, Zhang YY, Wei JQ, Han Y, Han L, Yang JP. A Comparative Study on Efficacy and Safety of Propofol versus Dexmedetomidine in Sleep Apnea Patients undergoing Drug-Induced Sleep Endoscopy: A CONSORT-Prospective, Randomized, Controlled Clinical Trial. Biomed Res Int. 2018 Nov 1;2018:8696510. doi: 10.1155/2018/8696510. eCollection 2018. PMID 30515416
- [Background] Kandil A, Subramanyam R, Hossain MM, Ishman S, Shott S, Tewari A, Mahmoud M. Comparison of the combination of dexmedetomidine and ketamine to propofol or propofol/sevoflurane for drug-induced sleep endoscopy in children. Paediatr Anaesth. 2016 Jul;26(7):742-51. doi: 10.1111/pan.12931. Epub 2016 May 23. PMID 27212000
- [Background] Gazzaz MJ, Isaac A, Anderson S, Alsufyani N, Alrajhi Y, El-Hakim H. Does drug-induced sleep endoscopy change the surgical decision in surgically naive non-syndromic children with snoring/sleep disordered breathing from the standard adenotonsillectomy? A retrospective cohort study. J Otolaryngol Head Neck Surg. 2017 Feb 13;46(1):12. doi: 10.1186/s40463-017-0190-6. PMID 28193298
- [Background] Baldassari CM, Lam DJ, Ishman SL, Chernobilsky B, Friedman NR, Giordano T, Lawlor C, Mitchell RB, Nardone H, Ruda J, Zalzal H, Deneal A, Dhepyasuwan N, Rosenfeld RM. Expert Consensus Statement: Pediatric Drug-Induced Sleep Endoscopy. Otolaryngol Head Neck Surg. 2021 Oct;165(4):578-591. doi: 10.1177/0194599820985000. Epub 2021 Jan 5. PMID 33400611